CLINICAL TRIAL: NCT00812929
Title: A Multi-centre, Randomized, Double-blind, Five-way Crossover Study Evaluating the Dose Response and Duration of Action of GSK2190915 Compared to Placebo in Subjects With Mild Asthma Who Experience Exercise Induced Bronchoconstriction.
Brief Title: A Clinical Trial to Test a Study Drug in Volunteers Who Develop Asthma Following Exercise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 112025
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Results first posted 2017-09-19 (Actual); Last update posted 2017-09-19 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Asthma, Exercise Induced Asthma, Exercise Induced Bronchospasm
MeSH Terms: conditions — Asthma; Asthma, Exercise-Induced | interventions — 3-(3-tert-butylsulfanyl-1-(4-(6-ethoxypyridin-3-yl)benzyl)-5-(5-methylpyridin-2-ylmethoxy)-1H-indol-2-yl)-2,2-dimethylpropionic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GSK2190915 10 mg (Experimental)
  Interventions: Drug: GSK2190915
- GSK2190915 50 mg (Experimental)
  Interventions: Drug: GSK2190915
- GSK2190915 100 mg (Experimental)
  Interventions: Drug: GSK2190915
- GSK2190915 200 mg (Experimental)
  Interventions: Drug: GSK2190915

INTERVENTIONS:
Drug: Placebo — The current study will include a placebo arm to allow for a valid evaluation of adverse events attributable to GSK2190915 versus those independent of GSK2190915.
  Arms: Placebo
Drug: GSK2190915 — This study will assess FEV1 at various intervals following exercise challenge in subjects who have been administered a single dose of 10 mg, 50 mg, 100 mg, or 200 mg GSK2190915, compared to a placebo control.
  Arms: GSK2190915 10 mg; GSK2190915 100 mg; GSK2190915 200 mg; GSK2190915 50 mg

SUMMARY:
This study is intended to determine the dose response and duration of action of GSK2190915 in mild asthmatic adult subjects who experience exercise-induced bronchoconstriction.

DETAILED DESCRIPTION:
This study is intended to determine the dose response and duration of action of GSK2190915 in mild asthmatic adult subjects who experience exercise-induced bronchoconstriction. Subjects will be invited to complete a screening visit, during which time exercise induced bronchoconstriction must be demonstrated, defined as a decrease between 20-40% in FEV1 compared to baseline immediately following exercise challenge. Eligible subjects will complete a randomized, double-blind, five-way crossover study. Subjects will be randomized to a single dose of either 10 mg, 50 mg, 100 mg, 200 mg GSK2190915, or placebo during each treatment period. Each treatment period will last 2 days and will include various assessments following exercise challenge at 2, 9.5, and 24 hours post dose. A minimum 7 day washout between treatment periods will be required. Regardless if a subject completes or prematurely withdraws from the study, a follow up visit will be completed 7-21 days following last dose.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 55 years inclusive.
* Female subjects must be of non childbearing potential including pre-menopausal females with documented hysterectomy or double oophorectomy or tubal ligation or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 40 pg/ml (<140 pmol/L) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy. Hormone replacement therapy (HRT) is permitted for post-menopausal females.
* Male subjects must agree to use one of the protocol outlined contraception methods. This criterion must be followed from the time of the first dose of study medication until 3 months after administration of last dose.
* Body weight greater than or equal to 50 kg and Body mass index within range of 18.5-35.0 kg/m2 inclusive.
* Pre-bronchodilator FEV1 >70% of predicted at screening.
* Exercise induced bronchoconstriction, as defined as a 20-40% decrease in FEV1 compared to baseline immediately following exercise challenge at screening.
* Current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit with a pack history of less than or equal to 10 pack years [number of pack years = (number of cigarettes per day/20) x number of years smoked]
* Has provided signed and dated written informed consent
* Is able to understand and comply with the protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

* Chronic use of inhaled corticosteroids (ICS) for the treatment of persistent asthma.
* Past or present disease, which as judged by the investigator or medical monitor, may affect the outcome of this study or the subject's safety. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, gastrointestinal disease, renal disease, haematological disease, neurological disease, endocrine disease or pulmonary disease (with the exception of asthma, but including chronic bronchitis, emphysema, bronchiectasis or pulmonary fibrosis).
* Treated for or diagnosed with clinical depression within six months of screening or has a history of significant psychiatric illness.
* Known history of hypertension or is hypertensive at screening which, in the opinion of the Investigator, deems the subject unfit to complete exercise challenge. Hypertension at screening is defined as persistent systolic BP >150 mmHg or diastolic BP > 90mmHg.
* Known history of gastrointestinal bleeding.
* Respiratory tract infection within 2 weeks prior to the first dose of study medication.
* Asthma exacerbations requiring treatment with oral corticosteroids: any exacerbations within 4 weeks of the screening visit or two or more exacerbations within 2 months of the screening visit or admittance to hospital for an asthma exacerbation within 6 months of the screening visit.
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest and/or hypoxic seizures.
* History of alcohol/drug abuse or dependence within 12 months of the study. Abuse of alcohol defined as an average weekly intake of >14 drinks/week for men or >7 drinks/week for women. One drink is equivalent to (12 g alcohol) = 5 ounces (150 ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Use of prescription or non-prescription drugs (including CYP 3A4 inhibitors and inducers, vitamins and dietary or herbal supplements), from 14 days before screening until the follow-up visit, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study. Inhaled beta-2 agonists and acetaminophen (up to 4 g per day) for the treatment of minor ailments, eg headache, are permitted. Hormone replacement therapy (HRT) is also permitted for post-menopausal females.
* Unable to washout the following protocol defined prohibited medications within the defined times:

Medication Exclusion Period Oral or injectable corticosteroids - No use within 5 weeks of the screening visit Inhaled, Intranasal and topical steroids - No use within 4 weeks of the screening visit Long acting beta-2 agonists - No use within 48 hours of an exercise challenge or dosing or lung function testing Short acting beta-2 agonists - No use within 6 hours of an exercise challenge or dosing or lung function testing

* Following exercise challenge during the screening visit, the subject experiences a greater than 40% fall in FEV1 compared to baseline.
* Following exercise challenge during the screening visit, the subject is not able to recover to at least 20% of baseline FEV1 following administration of short acting beta-2 agonists.
* Requires rescue medication before all lung function assessments are completed following the exercise challenge at screening
* Symptomatic with hay fever at screening or predicted to have symptomatic hayfever during the time of exercise challenge which, in the opinion of the Investigator, would interfere with the outcome of the study.
* Participation in a study with a new molecular entity during the previous 3 months or 5 half-lives (whichever is longer), or participation in a study without a new molecular entity during the previous month or 5 half-lives (whichever is longer), prior to the first dose of study medication.
* Undergoing allergen desensitisation therapy.
* There is a risk of subject non-compliance with study procedures.
* History of blood donation (500 mL) within 2 months of starting the clinical study.
* A screening QTc value of >450msec, PR interval outside the range 120 to 220msec or an ECG that is not suitable for QT measurements (e.g. poorly defined termination of the T-wave).
* Positive pregnancy test for females.
* Positive test for hepatitis C antibody or hepatitis B surface antigen.
* Positive test for HIV antibodies.
* Positive pre-study urine cotinine/ breath carbon monoxide test and or urine drug/urine alcohol screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids and Benzodiazepines.
* Has an affiliation with the Investigative Site. Participation of site personnel, or their spouses or children, is not allowed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2008-12-01; Primary Completion 2009-06-01 (Actual); Study Completion 2009-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Kent SE, Bentley JH, Miller D, Sterling R, Menendez R, Tarpay M, Pearlman DS, Norris V. The effect of GSK2190915, a 5-lipoxygenase-activating protein inhibitor, on exercise-induced bronchoconstriction. Allergy Asthma Proc. 2014 Mar-Apr;35(2):126-33. doi: 10.2500/aap.2014.35.3723. PMID 24717789
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 112025 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112025 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112025 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112025 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112025 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112025 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112025 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase IIa multi-center study conducted in the United States from 02 December 2008 to 15 July 2009.
Pre-assignment Details: A total of 47 participants were randomized in the study who underwent a screening visit of 28 days prior to first dose of study medication.
Groups:
- P/A/D/B/C: In this sequence participants received treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 1, treatment A of oral single dose of aqueous solution of 10 milligrams (mg) GSK2190915 on Day 1 of treatment period 2, treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 3, treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 4 and treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- A/B/P/C/D: In this sequence participants received treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 1, treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 2, treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 3, treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 4 and treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- B/C/A/D/P: In this sequence participants received treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 1, treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 2, treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 3, treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 4, treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- C/D/B/P/A: In this sequence participants received treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 1, treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 2, treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 3, treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 4, treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- D/P/C/A/B: In this sequence participants received treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 1, treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 2, treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 3, treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 4, treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- C/B/D/A/P: In this sequence participants received treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 1, treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 2, treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 3, treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 4, treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- D/C/P/B/A: In this sequence participants received treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 1, treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 2, treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 3, treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 4, treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- P/D/A/C/B: In this sequence participants received treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 1, treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 2, treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 3, treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 4, treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- A/P/B/D/C: In this sequence participants received treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 1, treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 2, treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 3, treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 4, treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
- B/A/C/P/D: In this sequence participants received treatment B of oral single dose of aqueous solution of 50 mg GSK2190915 on Day 1 of treatment period 1, treatment A of oral single dose of aqueous solution of 10 mg GSK2190915 on Day 1 of treatment period 2, treatment C of oral single dose of aqueous solution of 100 mg GSK2190915 on Day 1 of treatment period 3, treatment P of oral single dose of aqueous solution of matching placebo on Day 1 of treatment period 4, treatment D of oral single dose of aqueous solution of 200 mg GSK2190915 on Day 1 of treatment period 5. Each treatment periods were separated by a minimum 7 days washout period. Each treatment period included an exercise challenge at 2, 9.5, and 24 hours post dose and concluded on completion of the assessments following exercise challenge at 24 hours post dose.
Period: Treatment Period 1
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 4 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1 (7 Days)
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 5 | 4 | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2 (7 Days)
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 5
Completed | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Treatment Period 3
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 4
Completed | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3 (7 Days)
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 4 | 4
Completed | 5 | 4 | 4 | 4 | 5 | 4 | 5 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 4 | 4 | 5 | 4 | 5 | 5 | 4 | 4
Completed | 5 | 4 | 4 | 4 | 5 | 4 | 5 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 4 (7 Days)
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 4 | 4 | 5 | 4 | 5 | 5 | 4 | 4
Completed | 5 | 4 | 4 | 4 | 5 | 4 | 5 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 5
Arm/Group | P/A/D/B/C | A/B/P/C/D | B/C/A/D/P | C/D/B/P/A | D/P/C/A/B | C/B/D/A/P | D/C/P/B/A | P/D/A/C/B | A/P/B/D/C | B/A/C/P/D
Started | 5 | 4 | 4 | 4 | 5 | 4 | 5 | 5 | 4 | 4
Completed | 5 | 4 | 4 | 4 | 5 | 4 | 5 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Eligible participants completed five treatment periods (single dose 10 mg, 50 mg, 100 mg, 200 mg GSK2190915 oral solution, compared to placebo control which was administered on Day 1 of each treatment period). Each treatment period lasted 2 days, with a minimum 7 day washout period between each treatment periods.
Arm/Group | Total
Number analyzed (Participants) | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.4 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximal Percentage Change From Pre-exercise Baseline Forced Expiratory Volume in 1 Second (FEV1) to the Minimum FEV1 Collected Within 60 Minutes Following the Exercise Challenge at 24 Hours Post Dose
Description: FEV1 was recorded in triplicate, with participant encouraged to inhale fully despite any presence of chest tightness. For FEV1, a pre-challenge Baseline was defined for each challenge time point as maximum of triplicate measurements performed prior to challenge. The maximal percentage change within 60 minutes following exercise challenge was derived by taking minimum (i.e., most negative) percentage change in FEV1 over 5, 10, 15, 30, 45 and 60 minutes post challenge. Percent change FEV1 = 100*(FEV1 - Pre-challenge FEV1)/ Pre-challenge FEV1. If the exercise challenge was not completed successfully (i.e. heart rate maintained at >=80% of the predicted value for 6 minutes), FEV1 maximal percent change (0-60)was set to be missing. Analysis was performed using a mixed effects model, including period, treatment and covariates for predose FEV1. Estimates and 95% confidence intervals for treatment difference between each active dose and placebo for each challenge time point were calculated.
Time Frame: Baseline (pre dose) and 60 minutes following the exercise challenge at 24 hours post dose of each treatment period.
Population: The 'Efficacy Population' was defined as all participants who received at least one dose of study medication and are not major protocol violators.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Placebo: Eligible participants received Placebo matching GSK2190915 oral solution which was administered with 100 milliliter (mL) of water on Day 1 of each treatment period.
- GSK2190915 10 mg: Eligible participants received single dose 10 mg GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of each treatment period.
- GSK2190915 50 mg: Eligible participants received single dose 50 mg GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of each treatment period.
- GSK2190915 100 mg: Eligible participants received single dose 100 mg GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of each treatment period.
- GSK2190915 200 mg: Eligible participants received single dose 200 mg GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of each treatment period.
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 46 | 45 | 45
Percent change | -7.61 (1.326) | -6.33 (1.314) | -7.09 (1.307) | -7.28 (1.314) | -5.09 (1.315)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; Test type: Superiority; Mean Difference (Net) = 1.29, 95% CI 2-sided [-1.56 to 4.13], Standard Error of Mean 1.440
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 50 mg; Test type: Superiority; Mean Difference (Net) = 0.53, 95% CI 2-sided [-2.32 to 3.37], Standard Error of Mean 1.440
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 100 mg; Test type: Superiority; Mean Difference (Net) = 0.33, 95% CI 2-sided [-2.52 to 3.18], Standard Error of Mean 1.441
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 200 mg; Test type: Superiority; Mean Difference (Net) = 2.53, 95% CI 2-sided [-0.31 to 5.37], Standard Error of Mean 1.438

2. Secondary Outcome: Maximal Percentage Change From Pre-exercise Baseline FEV1 to the Minimum FEV1 Collected Within 60 Minutes Following the Exercise Challenge at 2 and 9.5 Hours Post Dose
Description: FEV1 was recorded in triplicate, with participant encouraged to inhale fully despite any presence of chest tightness. For FEV1, a pre-challenge Baseline was defined for each challenge time point as maximum of triplicate measurements performed prior to challenge. The maximal percentage change within 60 minutes following exercise challenge was derived by taking minimum percentage change in FEV1 over 5, 10, 15, 30, 45 and 60 minutes post challenge. Percent change FEV1 = 100*(FEV1 - Pre-challenge FEV1)/ Pre-challenge FEV1. If the exercise challenge was not completed successfully (i.e. heart rate maintained at >=80% of the predicted value for 6 minutes), the FEV1 maximal percent change (0-60)was set to be missing. Analysis was performed using a mixed effects model, including period, treatment and covariates for predose FEV1. Estimates and 95% confidence intervals for treatment difference between each active dose and placebo for each challenge time point were calculated.
Time Frame: Baseline (pre dose) and 60 minutes following the exercise challenge at 2 and 9.5 hours post dose of each treatment period.
Population: Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Groups:
- Placebo: Eligible participants received Placebo matching GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of each treatment period.
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 46 | 45 | 45
Percent change
  2 Hours | -15.55 (1.437) | -13.04 (1.424) | -12.95 (1.416) | -12.76 (1.424) | -9.25 (1.425)
  9.5 Hours | -8.45 (1.222) | -8.33 (1.212) | -7.69 (1.206) | -4.96 (1.213) | -6.18 (1.213)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; 2 Hours; Test type: Superiority; Mean Difference (Net) = 2.52, 95% CI 2-sided [-0.72 to 5.75], Standard Error of Mean 1.638
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 10 mg; 9.5 Hours; Test type: Superiority; Mean Difference (Net) = 0.12, 95% CI 2-sided [-2.34 to 2.58], Standard Error of Mean 1.247
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 50 mg; 2 Hours; Test type: Superiority; Mean Difference (Net) = 2.60, 95% CI 2-sided [-0.64 to 5.84], Standard Error of Mean 1.637
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 50 mg; 9.5 Hours; Test type: Superiority; Mean Difference (Net) = 0.76, 95% CI 2-sided [-1.70 to 3.22], Standard Error of Mean 1.247
Statistical Analysis 5: Comparison: Placebo vs GSK2190915 100 mg; 2 Hours; Test type: Superiority; Mean Difference (Net) = 2.79, 95% CI 2-sided [-0.45 to 6.03], Standard Error of Mean 1.639
Statistical Analysis 6: Comparison: Placebo vs GSK2190915 100 mg; 9.5 Hours; Test type: Superiority; Mean Difference (Net) = 3.49, 95% CI 2-sided [1.02 to 5.95], Standard Error of Mean 1.248
Statistical Analysis 7: Comparison: Placebo vs GSK2190915 200 mg; 2 Hours; Test type: Superiority; Mean Difference (Net) = 6.30, 95% CI 2-sided [3.06 to 9.54], Standard Error of Mean 1.637
Statistical Analysis 8: Comparison: Placebo vs GSK2190915 200 mg; 9.5 Hours; Test type: Superiority; Mean Difference (Net) = 2.27, 95% CI 2-sided [-0.19 to 4.73], Standard Error of Mean 1.245

3. Secondary Outcome: Weighted Mean (WM) for FEV1 Percentage Change From Baseline Recorded During 0 to 60 Minutes Following Exercise Challenge (FEV1 WM0-60)
Description: FEV1 was recorded in triplicate, with participant encouraged to inhale fully despite any presence of chest tightness. For FEV1, a pre-challenge Baseline was defined for each challenge time point as maximum of triplicate measurements performed prior to challenge.Weighted mean FEV1 percentage change recorded during 0-60 minutes post challenge was determined for each challenge, by dividing area under curve (AUC) for percent change from Baseline FEV1 measurements at 5, 10, 15, 30, 45 and 60 minutes post challenge by time interval. Actual times were used to determine time interval where available; otherwise planned relative time was used. If one or more FEV1 values were missing, AUC was calculated over time interval of available values. If intermittent values were missing over a participant's profile,it was assumed to be linear between 2 available values for calculation of AUC. Analysis was performed using a mixed effects model, including period, treatment and covariates for predose FEV1.
Time Frame: Baseline (pre dose) and 0 to 60 minutes following exercise challenge at 2, 9.5 and 24 hours post dose of each treatment period.
Population: Efficacy Population.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 46 | 45 | 45
Percent change
  2 Hours | -5.20 (0.936) | -4.26 (0.926) | -4.08 (0.920) | -3.69 (0.926) | -2.04 (0.927)
  9.5 Hours | -2.43 (0.757) | -2.36 (0.750) | -1.21 (0.745) | 0.87 (0.750) | -0.32 (0.750)
  24 Hours | -0.25 (0.755) | 0.65 (0.747) | -0.08 (0.742) | -0.35 (0.747) | 1.46 (0.748)
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; 2 Hours; Test type: Superiority; Mean Difference (Net) = 0.94, 95% CI 2-sided [-1.37 to 3.25], Standard Error of Mean 1.170 — Estimates and 95% confidence intervals for treatment difference between each active dose and placebo for each challenge time point were calculated
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 10 mg; 9.5 Hours; Test type: Superiority; Mean Difference (Net) = 0.07, 95% CI 2-sided [-1.66 to 1.80], Standard Error of Mean 0.878 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 10 mg; 24 Hours; Test type: Superiority; Mean Difference (Net) = 0.90, 95% CI 2-sided [-0.82 to 2.63], Standard Error of Mean 0.873 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 50 mg; 2 Hours; Test type: Superiority; Mean Difference (Net) = 1.12, 95% CI 2-sided [-1.19 to 3.43], Standard Error of Mean 1.169 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: Placebo vs GSK2190915 50 mg; 9.5 Hours; Test type: Superiority; Mean Difference (Net) = 1.22, 95% CI 2-sided [-0.51 to 2.95], Standard Error of Mean 0.878 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: Placebo vs GSK2190915 50 mg; 24 Hours; Test type: Superiority; Mean Difference (Net) = 0.18, 95% CI 2-sided [-1.55 to 1.90], Standard Error of Mean 0.873 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: Placebo vs GSK2190915 100 mg; 2 Hours; Test type: Superiority; Mean Difference (Net) = 1.51, 95% CI 2-sided [-0.80 to 3.82], Standard Error of Mean 1.171 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: Placebo vs GSK2190915 100 mg; 9.5 Hours; Test type: Superiority; Mean Difference (Net) = 3.30, 95% CI 2-sided [1.57 to 5.03], Standard Error of Mean 0.879 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: Placebo vs GSK2190915 100 mg; 24 Hours; Test type: Superiority; Mean Difference (Net) = -0.10, 95% CI 2-sided [-1.83 to 1.62], Standard Error of Mean 0.874 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: Placebo vs GSK2190915 200 mg; 2 Hours; Test type: Superiority; Mean Difference (Net) = 3.17, 95% CI 2-sided [0.86 to 5.48], Standard Error of Mean 1.169 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: Placebo vs GSK2190915 200 mg; 9.5 Hours; Test type: Superiority; Mean Difference (Net) = 2.11, 95% CI 2-sided [0.38 to 3.84], Standard Error of Mean 0.877 — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: Placebo vs GSK2190915 200 mg; 24 Hours; Test type: Superiority; Mean Difference (Net) = 1.72, 95% CI 2-sided [-0.00 to 3.44], Standard Error of Mean 0.872 — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Time to FEV1 Recovery to Within 5 Percent of Baseline Following Exercise Challenge
Description: The time from maximal percentage change in FEV1 to recovery to within 5% of pre challenge Baseline (in minutes) was derived using actual sampling times. Time to FEV1 recovery= [SAS date/time of recovery(a) FEV1 - SAS date/time of FEV1 Maximum % Change0-60] / 60, where "a" is earliest recorded FEV1 either above pre-challenge Baseline or within 5% below pre challenge Baseline. Any unscheduled FEV1 measurements taken after last scheduled post challenge measurement was considered when deriving this endpoint. A corresponding censoring variable was derived for analysis to indicate whether recovery to within 5% of pre-challenge Baseline was achieved. The censoring variable was set to 1 if recovery to within 5% of Baseline was achieved. If recovery was not evident from data collected, time to recovery was calculated using the date/time of the last available post challenge FEV1 assessment and censoring variable was set to zero. Analysis was performed using a Cox proportional hazards model.
Time Frame: 0 to 60 minutes following exercise challenge at 2, 9.5 and 24 hours post dose of each treatment period
Population: Efficacy Population.
Measure: Median (95% Confidence Interval); unit: Minutes
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 46 | 45 | 45
Minutes
  2 Hours | 24.5 [15.0 to 36.0] | 15.0 [10.0 to 30.0] | 18.0 [5.0 to 35.0] | 10.0 [5.0 to 16.0] | 5.0 [0.0 to 12.0]
  9.5 Hours | 5.0 [0.0 to 18.0] | 9.0 [0.0 to 25.0] | 5.0 [0.0 to 10.0] | 0.0 [0.0 to 5.0] | 0.0 [0.0 to 5.0]
  24 Hours | 5.0 [0.0 to 16.0] | 0.0 [0.0 to 5.0] | 2.5 [0.0 to 6.0] | 5.0 [0.0 to 5.0] | 0.0 [0.0 to 5.0]
Statistical Analysis 1: Comparison: Placebo vs GSK2190915 10 mg; 2 Hours; Test type: Superiority; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.71 to 2.21] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 2: Comparison: Placebo vs GSK2190915 10 mg; 9.5 Hours; Test type: Superiority; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.59 to 2.06] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 3: Comparison: Placebo vs GSK2190915 10 mg; 24 Hours; Test type: Superiority; Hazard Ratio (HR) = 1.78, 95% CI 2-sided [0.93 to 3.43] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 4: Comparison: Placebo vs GSK2190915 50 mg; 2 Hours; Test type: Superiority; Hazard Ratio (HR) = 1.42, 95% CI 2-sided [0.81 to 2.48] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 5: Comparison: Placebo vs GSK2190915 50 mg; 9.5 Hours; Test type: Superiority; Hazard Ratio (HR) = 1.93, 95% CI 2-sided [1.01 to 3.66] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 6: Comparison: Placebo vs GSK2190915 50 mg; 24 Hours; Test type: Superiority; Hazard Ratio (HR) = 1.67, 95% CI 2-sided [0.86 to 3.25] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 7: Comparison: Placebo vs GSK2190915 100 mg; 2 Hours; Test type: Superiority; Hazard Ratio (HR) = 2.09, 95% CI 2-sided [1.19 to 3.69] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 8: Comparison: Placebo vs GSK2190915 100 mg; 9.5 Hours; Test type: Superiority; Hazard Ratio (HR) = 5.49, 95% CI 2-sided [2.75 to 10.94] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 9: Comparison: Placebo vs GSK2190915 100 mg; 24 Hours; Test type: Superiority; Hazard Ratio (HR) = 1.91, 95% CI 2-sided [1.00 to 3.64] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 10: Comparison: Placebo vs GSK2190915 200 mg; 2 Hours; Test type: Superiority; Hazard Ratio (HR) = 3.60, 95% CI 2-sided [2.00 to 6.48] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 11: Comparison: Placebo vs GSK2190915 200 mg; 9.5 Hours; Test type: Superiority; Hazard Ratio (HR) = 2.03, 95% CI 2-sided [1.07 to 3.87] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo
Statistical Analysis 12: Comparison: Placebo vs GSK2190915 200 mg; 24 Hours; Test type: Superiority; Hazard Ratio (HR) = 6.07, 95% CI 2-sided [2.90 to 12.71] — Hazard ratio = ratio of likelihood of recovery at any time on active treatment vs placebo

5. Secondary Outcome: Number of Participants Using a Short Acting Beta-2 Agonist (Rescue Medication) During 0 to 90 Minutes Following Exercise Challenge
Description: Rescue medication was provided to participants at any time and it was strongly recommended for participants with a FEV1 decrease of at least 40% following exercise challenge compared to Baseline. Rescue medication was administered 0 to 90 minutes post exercise challenge. Statistical analysis was supposed to be performed using logistic regression, however, the data was too sparse to permit any formal statistical analysis.
Time Frame: 0 to 90 minutes following exercise challenge of each treatment period
Population: Efficacy Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 46 | 45 | 45
Participants
  2 Hours | 1 | 1 | 2 | 1 | 0
  9.5 Hours | 1 | 0 | 0 | 0 | 0
  24 Hours | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Assessment of Vital Signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: All participants rested for at least 10 minutes in the supine position prior to vital signs recordings. Vital signs Baseline values for SBP and DBP for each treatment period were calculated using the mean value of triplicate pre dose readings. Triplicate readings were taken at least five minutes apart. Assessment was performed at pre dose, 2 hours, 9.5 hours and 24 hours prior to exercise challenge.
Time Frame: Pre dose, 2 hours, 9.5 hours and 24 hours prior to exercise challenge of treatment period
Population: All Subjects Population was defined as all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Millimeters of mercury (mmHg)
  SBP, Mean Pre Dose | 118.8 (10.21) | 117.2 (10.45) | 117.6 (11.53) | 117.4 (11.49) | 118.1 (11.33)
  SBP, 2 Hours, Pre Exercise | 120.1 (10.50) | 119.8 (11.50) | 119.1 (10.48) | 119.4 (10.42) | 120.3 (11.32)
  SBP, 9.5 Hours, Pre Exercise | 119.4 (10.50) | 117.0 (8.69) | 120.5 (11.37) | 119.7 (10.58) | 118.4 (11.86)
  SBP, 24 Hours, Pre Exercise | 117.2 (11.62) | 116.9 (10.73) | 117.4 (9.93) | 117.5 (11.00) | 119.8 (11.50)
  DBP, Mean Pre Dose | 71.7 (7.37) | 71.9 (7.40) | 71.5 (7.59) | 71.6 (6.65) | 71.9 (6.62)
  DBP, 2 Hours, Pre Exercise | 71.1 (6.93) | 72.2 (6.09) | 71.3 (7.60) | 71.6 (7.76) | 72.2 (6.66)
  DBP, 9.5 Hours, Pre Exercise | 71.9 (6.05) | 70.5 (7.01) | 72.0 (7.65) | 71.2 (7.79) | 71.9 (7.71)
  DBP, 24 Hours, Pre Exercise | 71.1 (7.23) | 72.0 (7.84) | 72.2 (6.52) | 71.1 (8.25) | 72.9 (8.85)

7. Secondary Outcome: Assessment of Vital Signs: Heart Rate (HR)
Description: All participants rested for at least 10 minutes in the supine position prior to vital signs recordings. Vital signs Baseline values for HR for each treatment period were calculated using the mean value of triplicate pre dose readings. Triplicate readings were taken at least five minutes apart. Assessment was performed at pre dose, 2 hours, 9.5 hours and 24 hours prior to exercise challenge.
Time Frame: Pre dose, 2 hours, 9.5 hours and 24 hours prior to exercise challenge of each treatment period
Population: All Subjects Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Beats per minute
  Mean Pre Dose | 64.0 (9.20) | 63.0 (7.62) | 64.0 (7.78) | 63.6 (7.48) | 64.7 (8.38)
  2 Hours, Pre Exercise | 67.5 (8.78) | 66.2 (9.08) | 67.2 (8.51) | 66.8 (6.95) | 67.2 (8.98)
  9.5 Hours, Pre Exercise | 72.9 (11.35) | 69.4 (8.97) | 72.8 (9.16) | 72.3 (8.27) | 69.4 (9.46)
  24 Hours, Pre Excercise | 68.3 (10.90) | 65.7 (8.32) | 67.7 (8.75) | 65.9 (8.03) | 65.6 (9.31)

8. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: All participants rested for at least 10 minutes in the supine position prior to ECG recordings. ECG Baseline values for each treatment period was calculated using the mean value of triplicate pre dose readings. Triplicate readings were taken at least five minutes apart. Assessment was performed at pre dose, 2 hours, 9.5 hours, 24 hours prior to exercise challenge and 60 minutes following exercise challenge at 2 hours. Participants with not clinically significant (NCS) abnormal values were reported. Potential clinical importance range for the ECG parameters are as follows: absolute QTc interval >450 millisecond (msec), increase from Baseline QTc >60 msec, PR interval <110 and >220 msec and QRS interval <75 and >110 msec. No participants reported clinically significant abnormal values.
Time Frame: Pre dose, 2 hours, 9.5 hours and 24 hours prior to exercise challenge and 60 minutes following exercise challenge at 2 hours of each treatment period
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Participants
  Pre dose 1, Abnormal - NCS | 15 | 20 | 20 | 18 | 19
  Pre dose 2, Abnormal - NCS | 17 | 19 | 21 | 18 | 21
  Pre dose 3, Abnormal - NCS | 23 | 21 | 20 | 19 | 22
  2 Hours, Pre Exercise, Abnormal - NCS | 21 | 22 | 15 | 19 | 20
  2 Hours, 60 minutes, Abnormal - NCS | 15 | 21 | 17 | 19 | 20
  9.5 Hours, Pre exercise, Abnormal - NCS | 12 | 18 | 17 | 16 | 18
  24 Hours, Pre exercise, Abnormal - NCS | 16 | 22 | 19 | 18 | 20

9. Secondary Outcome: Assessment of Clinical Chemistry Parameters: Albumin, Total Protein
Description: Blood samples were collected for the assessment of clinical chemistry parameters for albumin and total protein at pre dose and 25 hours and 30 minutes. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram/liter (G/L)
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Gram/liter (G/L)
  Albumin, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Albumin, Pre dose 1 | 44.5000 (3.30961) | 44.9091 (2.60427) | 44.4894 (3.24956) | 44.8667 (2.54594) | 44.9778 (3.20148)
  Albumin, 25Hours 30minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Albumin, 25Hours 30minutes | 45.8140 (2.23879) | 45.4222 (3.08581) | 45.7021 (2.43091) | 45.9111 (2.16188) | 45.8444 (2.53122)
  Total protein, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Total protein, Pre dose 1 | 71.9 (5.32) | 72.5 (4.05) | 71.4 (5.11) | 71.6 (4.16) | 71.3 (4.78)
  Total protein, 25Hours 30minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Total protein, 25Hours 30minutes | 73.2 (4.00) | 72.9 (3.59) | 73.5 (3.97) | 72.6 (2.73) | 72.8 (3.72)

10. Secondary Outcome: Assessment of Clinical Chemistry Parameters: Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Gamma Glutamyl Transferase (GGT)
Description: Blood samples were collected for the assessment of clinical chemistry parameters for ALP, ALT, AST and GGT at pre dose and 25 hours and 30 minutes. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
International units per liter (IU/L)
  ALP, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  ALP, Pre dose 1 | 76.6 (26.15) | 75.5 (24.29) | 75.6 (25.64) | 74.6 (23.85) | 75.3 (22.69)
  ALP, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  ALP, 25 Hours 30 minutes | 75.3 (23.26) | 75.7 (23.75) | 76.9 (27.15) | 75.2 (23.71) | 75.8 (25.73)
  ALT, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  ALT, Pre dose 1 | 30.7 (19.09) | 30.1 (17.66) | 31.2 (18.97) | 32.2 (26.62) | 39.6 (71.33)
  ALT, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  ALT, 25 Hours 30 minutes | 31.7 (20.04) | 29.6 (16.08) | 32.4 (19.49) | 31.4 (23.34) | 38.5 (66.01)
  AST, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  AST, Pre dose 1 | 24.5 (13.29) | 24.0 (10.26) | 25.4 (14.81) | 24.6 (11.42) | 27.3 (31.46)
  AST, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  AST, 25 Hours 30 minutes | 24.0 (10.14) | 23.3 (8.82) | 27.3 (19.39) | 23.9 (9.72) | 26.9 (31.33)
  GGT, Pre dose 1: number analyzed (Participants) | 43 | 41 | 46 | 45 | 45
  GGT, Pre dose 1 | 29.8 (29.45) | 28.1 (21.98) | 31.5 (27.08) | 32.8 (39.54) | 30.3 (30.77)
  GGT, 2 5Hours 30 minutes: number analyzed (Participants) | 42 | 43 | 46 | 45 | 45
  GGT, 2 5Hours 30 minutes | 29.5 (25.87) | 27.7 (20.81) | 32.9 (29.08) | 32.8 (38.13) | 31.0 (31.83)

11. Secondary Outcome: Assessment of Clinical Chemistry Parameters: Direct Bilirubin, Total Bilirubin, Creatinine
Description: Blood samples were collected for the assessment of clinical chemistry parameters for direct bilirubin, total bilirubin and creatinine at pre dose and 25 hours and 30 minutes. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Micromoles per liter (µmol/L)
  Direct Bilirubin, Pre dose 1: number analyzed (Participants) | 42 | 44 | 46 | 45 | 45
  Direct Bilirubin, Pre dose 1 | 2.361 (1.8484) | 2.332 (1.4326) | 2.230 (1.8336) | 2.318 (1.6769) | 2.280 (2.1874)
  Direct Bilirubin, 25 Hours 30 minute: number analyzed (Participants) | 42 | 45 | 46 | 45 | 45
  Direct Bilirubin, 25 Hours 30 minute | 2.443 (1.8938) | 2.204 (1.2952) | 2.453 (2.3266) | 2.584 (1.8454) | 2.242 (1.9230)
  Total Bilirubin, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Total Bilirubin, Pre dose 1 | 10.804 (5.6386) | 11.348 (5.0173) | 11.060 (5.6473) | 11.438 (5.8652) | 11.134 (7.3966)
  Total Bilirubin, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Total Bilirubin, 25 Hours 30 minutes | 10.737 (5.3078) | 10.412 (4.8479) | 11.388 (6.1270) | 10.982 (5.8387) | 10.906 (6.4426)
  Creatinine, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Creatinine, Pre dose 1 | 83.96594 (18.34701) | 87.93791 (20.15153) | 86.23702 (13.21355) | 86.80880 (13.90414) | 85.96409 (14.50499)
  Creatinine, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Creatinine, 25 Hours 30 minutes | 85.83023 (14.40704) | 86.71058 (14.11612) | 87.91098 (13.81935) | 87.57493 (13.41632) | 87.57493 (14.84895)

12. Secondary Outcome: Assessment of Clinical Chemistry Parameters: Calcium, Chloride, Glucose, Potassium, Sodium, Urea/Blood Urea Nitrogen (BUN)
Description: Blood samples were collected for the assessment of clinical chemistry parameters for calcium, chloride, glucose, potassium, sodium and urea/BUN at pre dose and 25 hours and 30 minutes post dose. Participants had to fast for at least 8 hours prior to visit. Participants fasted for glucose blood sample. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimole per liter (mmol/L)
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Millimole per liter (mmol/L)
  Calcium, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Calcium, Pre dose 1 | 2.35494 (0.112125) | 2.36061 (0.107377) | 2.35910 (0.112041) | 2.35417 (0.109681) | 2.35084 (0.108088)
  Calcium, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Calcium, 25 Hours 30 minutes | 2.37605 (0.105831) | 2.38300 (0.110640) | 2.39308 (0.096186) | 2.38078 (0.091593) | 2.37136 (0.093348)
  Chloride, Pre dose 1: number analyzed (Participants) | 44 | 43 | 47 | 45 | 45
  Chloride, Pre dose 1 | 105.2 (1.92) | 105.1 (2.04) | 105.2 (2.07) | 105.0 (2.34) | 105.1 (2.42)
  Chloride, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Chloride, 25 Hours 30 minutes | 104.7 (2.36) | 105.4 (1.85) | 105.2 (2.28) | 104.8 (2.05) | 105.5 (2.29)
  Glucose, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Glucose, Pre dose 1 | 4.80162 (0.783522) | 4.73601 (0.804663) | 4.97937 (0.843434) | 4.88735 (0.770075) | 4.95273 (0.768704)
  Glucose, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Glucose, 25 Hours 30 minutes | 4.99203 (0.859137) | 4.96753 (0.892300) | 4.73370 (0.824460) | 5.02921 (1.004730) | 5.07855 (1.164605)
  Potassium, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Potassium, Pre dose 1 | 4.40 (0.328) | 4.40 (0.456) | 4.31 (0.386) | 4.29 (0.320) | 4.36 (0.422)
  Potassium, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Potassium, 25 Hours 30 minutes | 4.43 (0.342) | 4.51 (0.362) | 4.44 (0.374) | 4.44 (0.322) | 4.50 (0.333)
  Sodium, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Sodium, Pre dose 1 | 140.6 (2.16) | 140.9 (2.23) | 140.1 (2.17) | 139.9 (2.37) | 140.2 (1.87)
  Sodium, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 44
  Sodium, 25 Hours 30 minutes | 140.0 (2.13) | 140.6 (2.34) | 140.3 (2.18) | 139.6 (2.03) | 140.2 (2.14)
  Urea/BUN, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Urea/BUN, Pre dose 1 | 5.8175 (1.32593) | 5.6390 (1.56766) | 5.7652 (1.24779) | 5.7120 (1.25759) | 5.6565 (1.31601)
  Urea/BUN, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 47 | 45 | 45
  Urea/BUN, 25 Hours 30 minutes | 5.6539 (1.12605) | 5.5930 (1.11343) | 5.7424 (1.06537) | 5.8786 (1.09666) | 5.5771 (1.30126)

13. Secondary Outcome: Assessment of Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Total Neutrophils (TN) (ANC - Absolute Neutrophil Count), Platelet Count, White Blood Cell Count (WBC)
Description: Blood samples were collected for the assessment of hematology parameters for basophils, eosinophils, lymphocytes, monocytes, TN, platelet count, WBC at pre dose and 25 hours and 30 minutes post dose. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells x 10^9 per liter
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Cells x 10^9 per liter
  Basophils, Pre dose 1: number analyzed (Participants) | 18 | 18 | 17 | 18 | 18
  Basophils, Pre dose 1 | 0.0306 (0.01326) | 0.0281 (0.01065) | 0.0276 (0.01133) | 0.0316 (0.02112) | 0.0298 (0.01261)
  Basophils, 25 Hours 30 minutes: number analyzed (Participants) | 17 | 18 | 19 | 18 | 18
  Basophils, 25 Hours 30 minutes | 0.0242 (0.01064) | 0.0303 (0.00968) | 0.0333 (0.01805) | 0.0282 (0.00944) | 0.0252 (0.01171)
  Eosinophils, Pre dose 1: number analyzed (Participants) | 18 | 18 | 17 | 18 | 18
  Eosinophils, Pre dose 1 | 0.2638 (0.21459) | 0.2574 (0.20600) | 0.2392 (0.15458) | 0.2563 (0.21963) | 0.2166 (0.11200)
  Eosinophils, 25 Hours 30 minutes: number analyzed (Participants) | 17 | 18 | 19 | 18 | 18
  Eosinophils, 25 Hours 30 minutes | 0.2241 (0.15104) | 0.2610 (0.18803) | 0.2431 (0.15657) | 0.2271 (0.18567) | 0.1974 (0.10502)
  Lymphocyte, Pre dose 1: number analyzed (Participants) | 28 | 28 | 27 | 28 | 28
  Lymphocyte, Pre dose 1 | 2.2320 (0.62143) | 2.2139 (0.56983) | 2.3156 (0.56904) | 2.3581 (0.66985) | 2.1852 (0.69204)
  Lymphocyte, 25 Hours 30 minutes: number analyzed (Participants) | 27 | 28 | 29 | 28 | 28
  Lymphocyte, 25 Hours 30 minutes | 1.8281 (0.47068) | 1.8847 (0.55807) | 1.9052 (0.48399) | 1.8809 (0.49456) | 1.8677 (0.62646)
  Monocyte, Pre dose 1: number analyzed (Participants) | 18 | 18 | 17 | 18 | 18
  Monocyte, Pre dose 1 | 0.4673 (0.18438) | 0.4366 (0.11641) | 0.4799 (0.10725) | 0.4671 (0.11368) | 0.4307 (0.12690)
  Monocyte, 25 Hours 30 minutes: number analyzed (Participants) | 17 | 18 | 19 | 18 | 18
  Monocyte, 25 Hours 30 minutes | 0.3912 (0.09575) | 0.4289 (0.12575) | 0.4489 (0.13018) | 0.4190 (0.11797) | 0.4084 (0.15112)
  TN, Pre dose 1: number analyzed (Participants) | 28 | 28 | 27 | 28 | 28
  TN, Pre dose 1 | 3.4340 (0.98614) | 3.3645 (0.92934) | 3.4151 (0.96375) | 3.6047 (1.19442) | 3.5448 (1.05765)
  TN, 25 Hours 30 minutes: number analyzed (Participants) | 27 | 28 | 29 | 28 | 28
  TN, 25 Hours 30 minutes | 3.6062 (1.16759) | 3.6962 (0.92202) | 3.7720 (1.08800) | 3.7813 (1.26257) | 3.5289 (1.13473)
  Plateletcount, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Plateletcount, Pre dose 1 | 241.8 (58.19) | 238.0 (51.85) | 243.0 (47.46) | 240.1 (50.26) | 238.4 (49.15)
  Plateletcount, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 46 | 45 | 45
  Plateletcount, 25 Hours 30 minutes | 242.7 (55.97) | 239.0 (48.39) | 243.3 (46.73) | 240.5 (50.51) | 238.0 (52.59)
  WBC count, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  WBC count, Pre dose 1 | 6.69 (1.689) | 6.58 (1.638) | 6.77 (1.627) | 6.79 (1.726) | 6.50 (1.465)
  WBC count, 25 Hours 30 minutes: number analyzed (Participants) | 43 | 45 | 46 | 45 | 45
  WBC count, 25 Hours 30 minutes | 6.56 (1.708) | 6.56 (1.434) | 6.67 (1.605) | 6.75 (1.650) | 6.39 (1.681)

14. Secondary Outcome: Assessment of Hematology Parameters: Hemoglobin, Mean Corpuscle Hemoglobin Concentration (MCHC)
Description: Blood samples were collected for the assessment of hematology parameters for hemoglobin and MCHC at pre dose and 25 hours and 30 minutes post dose. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
G/L
  Hemoglobin, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Hemoglobin, Pre dose 1 | 152.0 (13.75) | 152.9 (13.00) | 151.3 (14.44) | 152.4 (12.95) | 151.3 (14.58)
  Hemoglobin, 25 hours 30 minutes: number analyzed (Participants) | 43 | 45 | 46 | 45 | 45
  Hemoglobin, 25 hours 30 minutes | 151.1 (12.84) | 151.9 (13.80) | 157.8 (45.11) | 151.3 (12.93) | 151.2 (13.41)
  MCHC, Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  MCHC, Pre dose 1 | 340.5 (8.55) | 339.3 (8.77) | 341.2 (8.35) | 340.0 (8.88) | 338.6 (9.40)
  MCHC, 25 hours 30 minutes: number analyzed (Participants) | 43 | 45 | 46 | 45 | 45
  MCHC, 25 hours 30 minutes | 340.2 (9.14) | 341.1 (7.43) | 340.4 (9.30) | 340.4 (9.05) | 339.8 (9.96)

15. Secondary Outcome: Assessment of Hematology Parameters: Hematocrit
Description: Blood samples were collected for the assessment of hematology parameters for hematocrit at pre dose and 25 hours and 30 minutes post dose. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Ratio
  Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Pre dose 1 | 0.4463 (0.03720) | 0.4503 (0.03423) | 0.4431 (0.03885) | 0.4480 (0.03265) | 0.4465 (0.03864)
  25 Hours 30 Minutes: number analyzed (Participants) | 43 | 45 | 46 | 45 | 45
  25 Hours 30 Minutes | 0.4440 (0.03186) | 0.4451 (0.03765) | 0.4453 (0.03375) | 0.4442 (0.03244) | 0.4448 (0.03628)

16. Secondary Outcome: Assessment of Hematology Parameters: Mean Corpuscle Hemoglobin (MCH)
Description: Blood samples were collected for the assessment of hematology parameter for MCH at pre dose and 25 hours and 30 minutes post dose. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Picograms
  Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Pre dose 1 | 30.27 (2.078) | 30.14 (2.122) | 30.30 (2.032) | 30.25 (2.024) | 30.14 (2.008)
  25 Hours 30 Minutes: number analyzed (Participants) | 43 | 45 | 46 | 45 | 45
  25 Hours 30 Minutes | 30.19 (2.157) | 30.20 (2.050) | 30.27 (2.076) | 30.18 (2.050) | 30.32 (2.102)

17. Secondary Outcome: Assessment of Hematology Parameters: Mean Corpuscle Volume (MCV)
Description: Blood samples were collected for the assessment of hematology parameter for MCV at pre dose and 25 hours and 30 minutes post dose. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Femtoliter
  Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Pre dose 1 | 88.85 (5.589) | 88.75 (5.500) | 88.80 (5.464) | 88.96 (5.673) | 89.06 (5.703)
  25 Hours 30 Minutes: number analyzed (Participants) | 43 | 45 | 46 | 45 | 45
  25 Hours 30 Minutes | 88.74 (6.116) | 88.57 (5.612) | 88.89 (5.696) | 88.69 (5.625) | 89.23 (5.730)

18. Secondary Outcome: Assessment of Hematology Parameters: Red Blood Cell Count (RBC)
Description: Blood samples were collected for the assessment of hematology parameter for RBC at pre dose and 25 hours and 30 minutes post dose. Participants had to fast for at least 8 hours prior to visit. During treatment periods, fasting continued until a light meal was allowed 1 hour post dose.
Time Frame: Pre dose and 25 hours and 30 minutes post dose of each treatment period
Population: All Subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells x 10^12 per liter
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Cells x 10^12 per liter
  Pre dose 1: number analyzed (Participants) | 44 | 44 | 47 | 45 | 45
  Pre dose 1 | 5.038 (0.4699) | 5.086 (0.4255) | 5.005 (0.4853) | 5.050 (0.4044) | 5.030 (0.4756)
  25 Hours 30 Minutes: number analyzed (Participants) | 43 | 45 | 46 | 45 | 45
  25 Hours 30 Minutes | 5.018 (0.3819) | 5.039 (0.4533) | 5.023 (0.4253) | 5.025 (0.4112) | 4.998 (0.4557)

19. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect and medically significant.
Time Frame: Up to follow up (7 to 21 days) following last dose
Population: All Subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 44 | 45 | 47 | 45 | 45
Participants
  Any AEs | 4 | 4 | 4 | 0 | 4
  Any SAEs | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Percentage Change From Baseline in Blood Leukotriene B4 (LTB4)
Description: Analysis LTB4 levels in the blood samples indicated the extent of LTB4 inhibition following administration of GSK2190915 compared to Baseline. Baseline was the pre dose value. Change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (pre dose) up to 24 Hours post dose of each treatment period
Population: Pharmacodynamics (PD) Population was defined as participants in the 'All Subjects' Population for whom a PD sample (blood or urine) was obtained and analyzed. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
Percent change
  2 Hours, Pre exercise: number analyzed (Participants) | 8 | 8 | 10 | 9 | 9
  2 Hours, Pre exercise | -37.32 [-57.8 to 241.4] | -29.32 [-78.4 to 125.3] | -87.65 [-99.6 to 78.9] | -97.98 [-99.7 to 25.9] | -98.43 [-100.0 to -55.9]
  9.5 Hours, Pre exercise | -14.82 [-74.6 to 239.4] | -23.43 [-93.4 to 31.1] | -87.74 [-98.4 to -23.0] | -96.53 [-99.4 to -45.2] | -99.78 [-100.0 to -95.0]
  24 Hours, Pre exercise | 12.59 [-57.2 to 235.1] | -9.56 [-83.3 to 167.9] | -84.49 [-96.7 to -36.3] | -70.00 [-97.8 to 209.4] | -98.75 [-99.8 to -64.9]

21. Secondary Outcome: Percentage Change From Baseline in Urine Leukotriene E4 (LTE4)
Description: Analysis of LTE4 levels in the urine samples indicated the extent of LTE4 inhibition following administration of GSK2190915 compared to Baseline. Baseline was the pre dose value. Change from Baseline was calculated by subtracting the Baseline values from the individual post-randomization values.
Time Frame: Baseline (pre dose) up to 24 Hours post dose of each treatment period
Population: PD Population. Only those participants available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
Percent change
  2 Hours, Pre exercise | -0.30 [-13.3 to 89.6] | -19.68 [-58.1 to 5.4] | -12.58 [-76.8 to 971.1] | -9.71 [-53.8 to 24.4] | -12.29 [-65.3 to 55.3]
  2 Hours, 1 Hour 30 Minutes post dose | 6.61 [-49.0 to 83.6] | -28.97 [-84.4 to 1.4] | -39.12 [-81.9 to 920.7] | -28.67 [-71.0 to 18.3] | -30.02 [-85.6 to 53.8]
  9.5 Hours, Pre exercise post dose | 0.82 [-42.4 to 37.9] | -52.76 [-86.0 to 0.3] | -66.74 [-86.4 to 629.8] | -59.85 [-98.2 to -23.1] | -70.43 [-87.7 to -27.3]
  9.5 Hours, 1 Hour 30 Minutes post dose | 0.96 [-49.0 to 88.5] | -45.05 [-89.3 to -15.9] | -61.86 [-86.6 to -0.3] | -63.67 [-83.5 to -42.1] | -81.03 [-94.4 to 5.8]
  24 Hours, Pre exercise post dose: number analyzed (Participants) | 8 | 9 | 9 | 9 | 9
  24 Hours, Pre exercise post dose | -14.04 [-50.3 to 24.1] | -29.26 [-82.6 to 21.3] | -70.37 [-88.7 to 24.9] | -72.55 [-99.5 to -5.7] | -77.07 [-99.1 to -34.2]

22. Secondary Outcome: Derived Pharmacokinetic (PK) Parameters for GSK2190915
Description: PK samples were supposed to be collected at 10 minutes prior to the exercise challenge at 2 hours, 9.5 hours and 24 hours.
Time Frame: Pre dose, 2 hours, 3.5 hours, 9.5 hours, 11 hours and 24 hours following exercise challenge of each treatment period
Population: PK Population was defined as participants in the 'All Subjects' Population for whom a PK sample was obtained and analyzed. Data was not collected for this outcome measure.
Arm/Group | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were collected up to follow up (up to 7 to 21 days following last dose).
Description: All Subjects Population was used.
Groups:
- Placebo: Eligible participants received Placebo matching GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of the treatment period.
- GSK2190915 10 mg: Eligible participants received single dose 10 mg GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of the treatment period.
- GSK2190915 50 mg: Eligible participants received single dose 50 mg GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of the treatment period.
- GSK2190915 100 mg: Eligible participants received single dose 100 mg GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of the treatment period.
- GSK2190915 200 mg: Eligible participants received single dose 200 mg GSK2190915 oral solution which was administered with 100 mL of water on Day 1 of the treatment period.
Arm/Group | Placebo | GSK2190915 10 mg | GSK2190915 50 mg | GSK2190915 100 mg | GSK2190915 200 mg
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/45 | 0/47 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/45 | 0/47 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 4/44 | 4/45 | 4/47 | 0/45 | 4/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=44) | GSK2190915 10 mg (N=45) | GSK2190915 50 mg (N=47) | GSK2190915 100 mg (N=45) | GSK2190915 200 mg (N=45)
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.